CLINICAL TRIAL: NCT01867151
Title: Effetto Della Dieta Priva di Glutine in Soggetti Con BMS
Brief Title: Effect of Gluten Free Diet in Patients With Burning Mouth Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Prof. Pier Mannuccio Mannucci, Scientific Director, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMS2013
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Burning Mouth Syndrome
Keywords: Burning Mouth Syndrome; Gluten; Gluten Free Diet
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gluten free diet (Experimental): BMS patients following a GFD
  Interventions: Dietary Supplement: Gluten Free Diet
- Normal Diet (Sham Comparator): Patients with BMS maintaing a normal diet
  Interventions: Dietary Supplement: Normal Diet

INTERVENTIONS:
Dietary Supplement: Gluten Free Diet
  Arms: Gluten free diet
Dietary Supplement: Normal Diet
  Arms: Normal Diet

SUMMARY:
Gluten free diet (GFD) is now being tested in patients affected by schizophrenia, autism and multiple sclerosis, making GFD a possible therapeutic weapon not only for celiac disease or gluten sensitivity. In this protocol we investigate the effect of GFD in patients affected by burning mouth syndrome (BMS), a disease of unknown origin characterized by oral and especially tongue burning sensation, deeply decreasing the quality of life of patients

ELIGIBILITY:
Inclusion Criteria:

-Primary BMS

Exclusion Criteria:

* Celiac Disease
* Psychiatric Disorders
* intestinal autoimmune diseases
* Ongoing cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-05 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
oral pain | 28 days
  oral pain will be evaluated by means of visual analogue scales

SECONDARY OUTCOMES:
Quality of Life | 28 days
  quality of life of patients with BMS will be evaluated by means of SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luca Elli, MD, Principal Investigator — Fondazione IRCCS Cà Granda
Locations (1):
- Fondazione IRCCS Ca' Granda, Milan, Italy, Italy